CLINICAL TRIAL: NCT01477554
Title: PRONTO: Obstetric and Neonatal Emergency Training Program: A Cluster-Randomized Trial to Measure Impact
Acronym: PRONTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Mexican National Institute for Women (Unknown); Mexican Center for Gender Equity and Reproductive Health (Unknown); Secretary for Women, Chiapas (Unknown); Secretary for Women, Mexico state (Unknown)
Responsible Party: Principal Investigator, Dilys Walker, Profesora Asociada C, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2-845-6519
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy Related Complications
Keywords: Women; Maternal morbidity; Maternal mortality; Perinatal mortality; Perinatal morbidity; Training; Obstetric Emergency; Medical team; Simulation
MeSH Terms: conditions — Maternal Death; Perinatal Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Hospitals randomized to the control arm do not receive any intervention.
- PRONTO training (Experimental): PRONTO training is delivered to medical teams at hospitals randomized to this arm.
  Interventions: Other: PRONTO training

INTERVENTIONS:
Other: PRONTO training — PRONTO is an intervention consisting of two training modules for medical professionals. Module 1 is delivered over 2-3 days, takes place in the hospital, and consists of high-fidelity, low-tech simulations. The curriculum employs elements of the Team STEPPS program to strengthen teamwork and leadership skills, and the use of effective communication techniques. The activities and simulations have clear objectives and use evidenced-based medical concepts. Module 2, the follow-up training, uses the same teaching methodology as Module 1 to reinforce teamwork, communication, and emergency response skills, and incorporates new topics such as preeclampsia /eclampsia, shoulder dystocia and pelvic presentation.
  Arms: PRONTO training

SUMMARY:
Rates and causes of maternal mortality in Mexico have dropped only slightly; thus, reaching the internationally established Millennium Development Milestones (MDM) is still a distant goal. A fundamental part of reducing maternal and infant mortality is ensuring an adequate and timely response to obstetric emergencies. PRONTO2: Obstetric and Neonatal Emergency Training Program is an innovative training strategy based on simulations designed to train hospital personnel to respond to obstetric emergencies. The objective of this study is to implement PRONTO2 in selected hospitals to measure the effectiveness of the intervention in influencing key behaviors in hospital practices, as well as measuring maternal and neonatal outcomes in intervention versus control hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals must be located in Guerrero, Chiapas, or Mexico states
* Number of deliveries and cesareans was between 500 and 3000 in 2009

Exclusion Criteria:

* Inaccessible by car

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Perinatal mortality | 12 months
  Assess perinatal mortality over the 12 month period following the training intervention

SECONDARY OUTCOMES:
Death rate from obstetric hemorrhage | 12 months
  Number of deaths from obstetric hemorrhage/total number of obstetric hemorrhages
Death rate from preeclampsia/eclampsia | 12 months
  Number of deaths from preeclampsia/eclampsia / totaly number of preeclampsia/eclampsia cases
Serious maternal complications | 12 months
  Assess the number of serious obstetric complications over 12 months following training intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dilys M Walker, MD, Principal Investigator — National Institute of Public Health Mexico

REFERENCES:
- [Derived] Fritz J, Lamadrid-Figueroa H, Angeles G, Montoya A, Walker D. Health providers pass knowledge and abilities acquired by training in obstetric emergencies to their peers: the average treatment on the treated effect of PRONTO on delivery attendance in Mexico. BMC Pregnancy Childbirth. 2018 Jun 15;18(1):232. doi: 10.1186/s12884-018-1872-4. PMID 29902983
- [Derived] Fritz J, Walker DM, Cohen S, Angeles G, Lamadrid-Figueroa H. Can a simulation-based training program impact the use of evidence based routine practices at birth? Results of a hospital-based cluster randomized trial in Mexico. PLoS One. 2017 Mar 20;12(3):e0172623. doi: 10.1371/journal.pone.0172623. eCollection 2017. PMID 28319122
- [Derived] Walker D, Cohen S, Fritz J, Olvera M, Lamadrid-Figueroa H, Cowan JG, Hernandez DG, Dettinger JC, Fahey JO. Team training in obstetric and neonatal emergencies using highly realistic simulation in Mexico: impact on process indicators. BMC Pregnancy Childbirth. 2014 Nov 20;14:367. doi: 10.1186/s12884-014-0367-1. PMID 25409895